CLINICAL TRIAL: NCT06023615
Title: Multifaceted Intervention to Improve Graft Outcome Disparities in African American Kidney Transplants (MITIGAAT)
Brief Title: MITIGAAT: Multifaceted Intervention to Improve Graft Outcome Disparities in African American Kidney Transplants
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, David J. Taber, Professor-Faculty, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00127666; 1R01DK134326-01A1 (NIH)
Record Dates: First submitted 2023-08-21; First posted 2023-09-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Medication Adherence; Medication Compliance
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): Usual Care + mHealth/Telehealth
  Interventions: Other: mHealth app/dashboard
- Control Group (No Intervention): Usual Care + Attention Control

INTERVENTIONS:
Other: mHealth app/dashboard — In the interventional group, the subject would receive the standard care that is provided to all post-transplant kidney recipients plus an additional remote monitoring system and follow-up by utilizing an app known as the mHealth app/dashboard. This app is integrated with home-based monitoring of blood pressures, glucoses, and pharmacist-led scheduled televisits.
  Arms: Intervention Group

SUMMARY:
This is a randomized study to test a smartphone app that a pharmacist will use to help kidney transplant patients track their medications, blood pressures, and blood sugars in those with diabetes. The goal of this study is to improve care and outcomes in kidney transplant patients and, in particular, help African American patients have better outcomes after transplant.

DETAILED DESCRIPTION:
The overarching hypothesis for MITIGAAT is that late non-adherence and suboptimal control of diabetes and hypertension are more common in African American kidney recipients and are major contributors to health disparities. A multimodal intervention that addresses these issues will significantly reduce disparities. This hypothesis will be tested through a rigorously conducted, prospective, 2-year randomized controlled trial in 190 kidney transplant recipients from MUSC, designed to assess the following aims:

Aim 1. Determine the impact of this multilevel health services intervention on achieving improved adherence to tacrolimus, measured using tacrolimus trough variability and time in range in the treatment vs control arm.

Aim 2. Determine the impact of this multilevel health services intervention on blood pressure (BP) and glucose control (in those with DM) in the treatment vs control arm.

Aim 3. Conduct a cost-benefit analysis (CBA), assessing the estimated hospitalization and ED visit costs in the intervention arm vs the control arm and compare this to the costs needed to deliver the intervention.

Aim 4. Compare the incidence of acute rejection, graft loss and death in the intervention patients vs. a large contemporary national cohort of Veteran kidney transplant recipients while also assessing racial disparities for these health outcomes

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* ≥2 years post-kidney transplant

Exclusion Criteria:

* Non-kidney transplant recipient (liver, lung, heart, intestine, pancreas, bone marrow)
* Not capable of measuring own BP and glucose in those with diabetes
* Not capable of using mobile health application after adequate training
* Not capable of speaking, hearing, and reading English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Medication Adherence | 2 Years
  Medication adherence will be measured by using tacrolimus trough concentration variability, which is a validated proxy measure of medication adherence. This is defined as the intrapatient tacrolimus concentration coefficient of variation (CV): standard deviation divided by the mean for each patient. All outpatient true trough tacrolimus levels drawn will be used to calculate the tacrolimus CV. This will be assessed every 3 months, which aligns with the minimum lab draw schedule for kidney transplant recipients at out center. This will be analyzed using repeated measures methodology, estimating efficacy effect size using the time*treatment interaction term and disparity using the time*treatment*race interaction term.
Blood Pressure | 2 Years
  Blood pressure control will be defined as the mean of all systolic BPs checked by patients at home and the transplant center (ambulatory measures). Patients with a mean of SBP ≤140 mmHg will be considered controlled. We will aggregate and assess blood pressure levels every month (25 total); analyzed using repeated measures (time*treatment and disparity using the time*treatment*race interaction term).
Glucose Control | 2 Years
  Glucose control is defined as the mean measure of all glucoses (random or fasting). Those with DM and a mean random glucose ≤160 mg/dL will be considered to controlled. We will aggregate and assess glucose levels every month (25 total); analyzed using repeated measures (time*treatment and disparity using the time*treatment*race interaction term).
Cost-Benefit Analysis | 2 Years
  Conduct a cost-benefit analysis (CBA), assessing the estimated hospitalization and ED visit costs in the intervention arm vs the control arm and compare this to the costs needed to deliver the intervention.
Acute Rejection | 2 Years
  This is defined as the proportion of patients in each arm with a renal allograft biopsy showing at least grade 1A rejection by Banff criteria. Per usual care practices, all patients are required to have biopsy confirmation of rejection episodes within 24 hours of onset of treatment for acute rejection. It is standard care that all kidney allograft biopsies performed for transplant recipients occur at the transplant center (study institution). Biopsies will be read by a blinded local pathologist, as usual care. This will be assessed using time to event analyses..
Graft Failure | 2 Years
  This is defined as the proportion of patients in each arm with graft failure, which is a composite outcome of either return to chronic dialysis, nephrectomy, re-transplant, or death. The timing and cause of each graft loss will be recorded for comparative analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Overstreet M, Culpepper H, DeHoff D, Gebregziabher M, Posadas Salas MA, Su Z, Chandler J, Bartlett F, Dunton P, Carcella T, Taber D. Multifaceted Intervention to Improve Graft Outcome Disparities in African American Kidney Transplants (MITIGAAT Study): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Oct 10;13:e57784. doi: 10.2196/57784. PMID 39388231